CLINICAL TRIAL: NCT05602909
Title: Evaluation of the Efficiency of Guided Biaxial Alveolar Distraction Device in Posterior Atrophic Mandible (A Clinical Trial)
Brief Title: Guided Biaxial Alveolar Distraction Device in Posterior Atrophic Mandible
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Distractors_2022
Record Dates: First submitted 2022-10-14; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Mandible; Deformity
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guided biaxial distraction (Experimental)
  Interventions: Device: Guided biaxial alveolar distraction device

INTERVENTIONS:
Device: Guided biaxial alveolar distraction device — A crestal incision will be done, a surgical guide will be placed to assist the correct position of osteotomy, an Extraosseous alveolar distractor will be placed on the ridge to mark screw sites and then will be removed, A distractor will be stabilized to the basal segment with a monocortical screw.

SUMMARY:
Atrophic alveolar bone presents a unique difficulty, preventing correct implant placement and affecting long-term results. There are different techniques that are recommended to restore the proper length of the posterior ridge of the mandible and thus achieve proper form and function, one of those is distraction osteogenesis. Refinements in the technique of distraction can improve the treatment outcome and decrease postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the posterior atrophic mandible.
* The distance from the alveolar crest to the upper border of the canal is not less than 5 mm.
* Adult patients from 30-60 years old with no gender predilection who agreed to present for follow-up visits for a minimum postoperative period of 4 months.
* Patientswithanadequateoralhygiene.
* The patient should be psychologically accepting of the involved procedures.

Exclusion Criteria:

* Medically compromised patients contradicting operation (ASA III, IV & V).
* Patients receiving radiotherapy or chemotherapy or bisphosphonate.
* Bonediseases(Osteoporosis,Osteopetrosis,Osteomalacia...etc.)
* Any habits that might retard healing such as heavy smoking and alcoholism.
* A history of any grafting procedure at the designated area.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain scorre | at 1, 7 and 14 days
  It will be assessed on daily basis for one week through a 10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
change in wound healing | at 1, 7 and 14 days
  The sutured wounds will be examined for wound dehiscence as (Yes for present and No for absent)
Change in mental nerve reflex | Baseline, after 2 weeks and 1 month
  Mental nerve blink reflex responses to electrical stimuli given with a small bipolar pediatric stimulating electrode to the center of the mental nerve distribution on the chin and lower lip on each side will be recorded bilaterally with surface electrodes on the orbicularis oculi muscles with Viking IV EMG equipment
Change in bone density | Baseline,1 month, 3 months
  Bone density at the distracted area, the length will be gained and displacement of transported segment lingually will be evaluated using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt